CLINICAL TRIAL: NCT01119326
Title: A Phase I/II Study of Autologous Fat Transfer for Scar Prevention and Remodeling
Brief Title: Autologous Fat Transfer for Scar Prevention and Remodeling
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 503-2012
Record Dates: First submitted 2010-04-27; First posted 2010-05-07 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Wound
Keywords: scar prevention; healing; tissue; AFT; scar analysis
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo procedure
  Interventions: Procedure: Autologous Fat Transfer
- Autologous Fat Transfer (AFT) group (Experimental): Subjects will be registered in the context of either the Early AFT subgroup, or the Delayed AFT subgroup based on the timing of their wound closure: early AFT subgroup will contain subjects who are medically stable such that study sites are amenable to AFT within 2-4 weeks of definitive closure (STSG) or healing (secondary closure) and the delayed AFT subgroup will contain subjects who are medically stable such that study sites are amenable to AFT within 6 months or more of definitive closure (STSG) or healing (secondary closure
  Interventions: Procedure: Autologous Fat Transfer

INTERVENTIONS:
Procedure: Autologous Fat Transfer — one site will be treated with AFT For placebo treated (control) sites, an equal number of empty cannula passes will be administered using a similar technique described for the AFT.

SUMMARY:
The purpose of this research study is to find out if it is safe and feasible to improve the appearance and quality of a scar by using a procedure in which adipose tissue (fat) is taken from other parts of your body and injected, or transplanted into a scar. This procedure is called autologous fat transfer (AFT). The main goal of this study is to see if AFT is safe and can improve the quality and appearance of scar tissue. Another main goal is to determine how much tissue should be transplanted to get the best results.

DETAILED DESCRIPTION:
Before you begin study treatment, you will have the following tests and procedures:

* A physical examination
* A review of your medical history. You will be asked about any history of psychiatric illness.
* You will be asked about any medications you might be currently taking. In addition, you will be asked about alcohol and drug use.
* Pregnancy test, if you are a woman of childbearing potential.
* Digital photography of the treatment sites.
* Scar assessment - you will be asked to complete a quick and simple questionnaire about the appearance of your scars and how well they are healing/have healed.
* Passive and Active range of motion assessment (P/AROM) - If your study scars extend over a joint such as the elbow, or a finger knuckle, you will be tested to see how well you can move or bend the joint before and after the study treatment.
* After screening, but prior to AFT procedure, you may need to undergo additional tests. These tests may include further laboratory assessments, a chest x-ray, or electrocardiogram (ECG). The requirement for the additional testing is largely depending on your age, recent surgical or medical history, or a medical condition indicating the need for these tests.
* Outpatient surgery procedure that will include anesthesia that puts you to sleep (either with or without a breathing tube), medicines given through an IV (into your veins), and/or local numbing medicine, such as lidocaine. You will receive ALL of the usual standard monitoring, medications, safety precautions, and care that is provided for any patient undergoing any surgery, including antibiotics as needed, pain medicine as needed (during and after your procedure) and other supportive care as needed.
* You will have 2 treatment sites identified for AFT in this study. Under anesthesia, you will have skin biopsies for research purposes only taken prior to study procedures from each designated treatment area. Both treatment sites will be similar in size and location on your body. One of these sites will be treated using the AFT procedure; the other will be treated using a fake procedure (placebo procedure).
* The surgeon will remove fat tissue from under you skin using standard liposuction methods.
* This tissue will be washed and concentrated to remove unwanted fluids and medicines and then injected under the designated skin grafts/scars using a small needle.
* There will be follow-up visits done 1 week, 1 month, 3 months, 6 months, and 12 months after the AFT procedure to perform the following tests and procedures:
* A physical examination
* A review of your medical history
* You will be asked about any medications you might be currently taking
* Digital photography of the treatment sites.
* Scar assessment - you will be asked to complete a questionnaire about the appearance of your scars and how well they are healing.
* Active range of motion assessment (AROM) - If your site spans a joint, you will be tested to see how well you can move the joint.
* As part of this research study, two skin biopsies will be taken from each study site (at time of treatment, 6 months, and 12 months after AFT procedure only). A skin biopsy is a routine procedure which involves obtaining a very small skin sample (2-4 mm) with a special instrument (punch biopsy) that cuts out a small circular piece of skin. If needed, the area where the biopsy was taken may be closed with stitches.

ELIGIBILITY:
Inclusion Criteria:

1. At least 2 separate (i.e. non-contiguous) wounds/scars previously healed by placement of a STSG and/or by secondary intention ("study sites"), each ≤ 50cm2 in size (area).

   o The study sites should be similar in size and anatomical location (e.g. upper arms; trunk; legs) to the extent practically possible
2. Adequate adipose depot for tissue harvest
3. For Early AFT Subgroup:

   o medically stable such that study sites are amenable to AFT within 2-4 weeks after definitive closure(STSG) or healing (secondary closure)

   For Delayed AFT Subgroup:

   o medically stable such that study sites are amenable to AFT at least 6 months after definitive closure(STSG) or healing (secondary closure)
4. Age range: 18-65 years
5. Negative pregnancy test
6. Able and willing to provide verbal and written informed consent.
7. Subject should begin protocol initiation within 2 weeks of being enrolled.

Exclusion Criteria:

1. Sepsis
2. Life or limb-threatening injury/disease
3. Prior history of non-compliance
4. Active drug use/abuse
5. Active psychiatric illness
6. Pregnancy
7. Active cancer, or new diagnosis of cancer within the past 5 years, with the exception of basal cell and squamous cell carcinomas, as long as the subject is disease free at the time of enrollment and that the previous diagnosis was not at a site to be treated by AFT.
8. History of bleeding tendency/inability to clot, and/or International normalized ratio(INR) ≥ 2.2
9. Life-threatening allergic reaction to one of the medications/agents to be used in the study with no acceptable alternative/substitute identifiable
10. Use of steroid injections, pressure garments, silicone sheeting or other similar scar management modalities and cannot be discontinued during study participation.
11. Incarceration.
12. Active duty military personnel (at UF site only)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-04; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
To determine the safety and feasibility of using AFT in early and delayed treatment settings to positively enhance the quality and appearance of overlying scar and to determine the safety and impact of AFT "dose" on scar quality and appearance. | 4 times for a year
  If no Dose Limiting Toxicity (DLT) is observed ,dose escalation will occur. Study sites/scars will be delineated by tracings, digital photography,scar assessment scale,and measures of scar elasticity and color. To correlate efficacy with graft quality, a sample of each adipose harvest will be sent to the laboratory for quantitative analysis of the stromal vascular fraction (SVF) with the adipose sample.

SECONDARY OUTCOMES:
To determine the correlation of subjective and objective scar assessment tools for serial, prospective scar analysis. | 4 times for a year

CONTACTS AND LOCATIONS:
Overall Officials: Adam Katz, MD, Principal Investigator — University of Florida
Locations (3):
- United States (3):
  - University of Florida, Gainesville, Florida
  - Institute of Surgical Research (ISR)/Brooke Army Medical Center (BAMC), Fort Sam Houston, Texas
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No